CLINICAL TRIAL: NCT03843723
Title: Exercise Pulse Oximetry and Pre-flight Evaluation of Adult Cystic Fibrosis (CF) Patients
Brief Title: Cystic Fibrosis and Fit-to-Fly
Acronym: CyFF
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: The Norwegian Resouce Centre for Cystic Fibrosis (Unknown); Norwegian National Adivisory Unit on Rare Disorders (Unknown); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Aina Akerø, Principal Investigator, MD PhD, Oslo University Hospital
Other Study IDs: 2018/1607 (REK)
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis; Hypoxemia; Lung Diseases
Keywords: Pre-flight evaluation; Air travel; Pulseoximetry; Exercise desaturation; Hypobaria; Hypoxemia
MeSH Terms: conditions — Cystic Fibrosis; Hypoxia; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pre-flight evaluation — All the participants receive the interventions as part of their routine medical care during their annual visit for CF follow-up. Oxygen saturation are measured by pulse oximetry. Exercise testing is performed by 6MWT and CPET. Pre-flight evaluation is performed by HAST.

SUMMARY:
Due to the hypobaric hypoxia during air travel, some patients with Cystic Fibrosis (CF) need supplemental oxygen during air travel.

The study aims to evaluate if adding exercise desaturation to the pre-flight evaluation will help predict requirements for in-flight supplemental oxygen.

DETAILED DESCRIPTION:
According to the British Thoracic Society (BTS) recommendations regarding pre-flight evaluation in patients with pulmonary disease, pre-flight arterial oxygen saturation or lung function tests do not discriminate sufficiently between those who need supplemental oxygen during flights, and those who can do without.Therefore, more extensively use of Hypoxia Altitude Simulation test (HAST) has been advocated. However, this test is not widely available. Previous studies have shown that exercise testing is useful for the prediction of in-flight hypoxemia. The investigators have previously developed a pre-flight algorithm for patients with chronic obstructive pulmonary disease (COPD), based on oxygen saturation measured by pulse oximetry at rest and during exercise (six minute walking test (6MWT)). It remains unknown as to whether these results are applicable to the CF population.

The current study aims to validate the pre-flight algorithm for patients with CF. Since a maximum cardiopulmonary exercise test (CPET) is recommended in the routine CF-control, the investigators also aim to evaluate whether the use of CPET predicts in-flight hypoxemia with greater accuracy than 6MWT, and whether CPET may replace HAST.

ELIGIBILITY:
Inclusion Criteria:

* Adult CF patients (age from 18 years)
* Signed informed consent

Exclusion Criteria:

* Ongoing exacerbation
* Unable to fulfill a CPET or 6MWT
* Long-term oxygen treatment (LTOT)
* Severe heart disease
* Language problems that interfere with data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with CF evaluated at the Norwegian Resource Centre for Cystic Fibrosis at the Dep. of Pulm. Med. Oslo University Hospital
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Does oxygen saturation during exercise predict in-flight hypoxemia in adult patients with CF? | 1 day
  Oxygen saturation is measured by pulse oximetry (SpO2) during exercise and HAST

CONTACTS AND LOCATIONS:
Overall Officials: Aina Akerø, MD PhD, Principal Investigator — Oslo University Hospital, Dept. of Pulm. Med.
Locations (1):
- Oslo University Hospital Ullevaal, Department of Pulmonary Medicine, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participants data available to other researchers due to restrictions from Oslo University Hospital

REFERENCES:
- [Background] Edvardsen A, Akero A, Christensen CC, Ryg M, Skjonsberg OH. Air travel and chronic obstructive pulmonary disease: a new algorithm for pre-flight evaluation. Thorax. 2012 Nov;67(11):964-9. doi: 10.1136/thoraxjnl-2012-201855. Epub 2012 Jul 5. PMID 22767877
- [Background] Ahmedzai S, Balfour-Lynn IM, Bewick T, Buchdahl R, Coker RK, Cummin AR, Gradwell DP, Howard L, Innes JA, Johnson AO, Lim E, Lim WS, McKinlay KP, Partridge MR, Popplestone M, Pozniak A, Robson A, Shovlin CL, Shrikrishna D, Simonds A, Tait P, Thomas M; British Thoracic Society Standards of Care Committee. Managing passengers with stable respiratory disease planning air travel: British Thoracic Society recommendations. Thorax. 2011 Sep;66 Suppl 1:i1-30. doi: 10.1136/thoraxjnl-2011-200295. No abstract available. PMID 21856702
- [Derived] Akero A, Edvardsen E, Finstad PL, Skrede B, Osterhaug M, Backman S, Edvardsen A, Skjonsberg OH. Air travel and cystic fibrosis: An algorithm to assess the risk of In-Flight Hypoxemia. J Cyst Fibros. 2025 Sep;24(5):963-969. doi: 10.1016/j.jcf.2025.05.004. Epub 2025 Jun 3. PMID 40467430